CLINICAL TRIAL: NCT04379960
Title: Identification of Immunogenic Neo-epitopes for the Development of Personalised Pancreatic Cancer Vaccines
Acronym: CanVac
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/LO/1512
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2016-09

CONDITIONS: The Initial Aim of This Project is to Perform in Vitro Validation of Neoepitope Candidates Selected From Available Mutanome Data
MeSH Terms: interventions — Peptides

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human blood from healthy donors, who donate blood at the Blood Donation Centres.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Peptides: PBMCs will be incubated with peptides.
  Interventions: Other: Peptides
- W/o peptides: PBMCs will be incubated without peptides.
  Interventions: Other: Peptides

INTERVENTIONS:
Other: Peptides — Peptides will be added to PBMCs in in vitro cell culture.

SUMMARY:
Human pancreatic cancer has a very poor prognosis with an overall survival rate of less than 5%. Current treatment regimens are ineffective and even if the patient responds to initial treatments, relapse is common due to the survival of small populations of resistant cancer cells.

The immune system is capable of recognising and eliminating invading organisms by virtue of differences in their appearance when compared to normal components of the body. Cancer cells also have a different appearance compared to normal cells. However, these differences are often too small and weak to stimulate the immune system sufficiently to respond effectively to eliminate the tumour.

Our aim is to analyse the small differences between healthy and cancer cells in pancreatic cancer patients. Analysis of the genetic information from 100 pancreatic cancer patients has allowed us to design molecules that display each of these small differences. We now intend to analyse each of these, with respect to their ability to stimulate an immune response against cancer. We then intend to take all validated molecules and incorporate them into vaccines carried by viral vectors. These vaccines can be used to train the patient's immune system to respond more effectively when it encounters these particular differences in the patient's body and thus mount an efficient attack on the cancer cells specifically.

Surplus material from blood donations will be used to isolate individual components of the immune system, which can be examined for their response to these altered molecules in the laboratory. On completion of this project, we will have viral vaccine libraries that can be tested in future research projects. Ultimately, we hope to transfer this regime to the clinic by selecting an appropriate viral vaccine library to deliver as a personalised therapeutic that can eliminate cancer and prevent cancer recurrence within each patient.

DETAILED DESCRIPTION:
Background Pancreatic ductal adenocarcinoma (PDAC) is one of the most aggressive tumour types, with an extremely poor prognosis. Without active treatment, patients with metastatic PDAC have a mean survival of 3-5 months [1]. Current advances in surgical and adjuvant treatments have failed to improve overall survival rates since the 1970s. Thus, new treatment strategies, that are not cross resistant with conventional chemotherapy-based regimes are imperative. Recently, attention in cancer therapy has focused more heavily on immune-based strategies as these therapies act through a mechanism that is distinct from chemotherapy or radiation therapy and represent a non-cross-resistant treatment option [2]. Immune based therapies aim to stimulate robust T cell responses against tumour antigens. However, significant challenges exist in the development of these regimes. These include poor immunogenicity of the tumours and the presence of a highly immunosuppressive environment within the tumour [3, 4]. The clinical potential of various tumour vaccination strategies has been demonstrated in early phase clinical trials, with some promising immunological and clinical responses in PDAC patients [5-8]. A number of hurdles still need to be overcome in the development of an ideal PDAC vaccine. Crucially, specific tumour antigens must be identified that elicit a strong and specific immune response as failure of past cancer vaccine trials can be attributed in large part to selection of inappropriate tumour antigens that have weak inherent immune potential [9, 10]. Current advances in high throughput profiling technologies as enabled rapid determination of the genomic states of cancer cells such that comprehensive data regarding individual mutanomes is now available [11, 12]. It is also now possible to select missense mutations identified through the exome sequencing on the basis of their HLA binding capacity for production of synthetic peptides that can be presented by a desired HLA molecule [12, 13]. The development of this platform has allowed us to analysed published data from 100 PDAC patients [14] and establish a dataset containing high-affinity HLA-A2 and HLA-DP4 (the most abundant HLA class I and II molecules [15, 16]) and HLA-E*01:01 and HLA-E*01:03-restricted neo-epitopes for analysis as peptide vaccine candidates.

Hypothesis Sequence analysis has allowed us to develop a peptide library of neo-epitopes that are expressed at high frequency in patient populations and have high binding affinities compared to their wild-type counterpart to HLA-A2, HLA-DP4, HLA-E*01:01 or HLA-*01:03 molecules. We hypothesise that a number of these will be sufficiently immunogenic to stimulate a T cell interferon-γ (IFN-γ) response in vitro, that will translate to an in vivo anti-tumour response. Immunogenic neo-epitopes can then be combined in a peptide vaccination program using adjuvants such as oncolytic viruses for targeted delivery and expression within tumours of PDAC patients to stimulate robust and long-term anti-tumour responses.

Aim The initial aim of this project is to perform in vitro validation of neo-epitope candidates selected from available mutanome data to determine their immunogenicity using peripheral blood mononuclear cells (PBMCs) from healthy individuals.

Research Plan PBMC samples from healthy individuals will be HLA typed using commercially available reagents from thermofisher scientific. HLA-A2, HLA-DP4, HLA-E*01:01 and/or HLA-E*01:03 positive samples will be pulsed with peptides selected after bioinformatics analysis of available sequence data. IFN-γ and interleukin-2 (IL-2) production by the T cells in the samples will be evaluated by ELISA after two rounds of stimulation within a two weeks time as a measure of peptide immunogenicity. Once immunogenic peptides have been identified, their wild-type counterparts will be analysed in parallel to confirm specificity for the mutated epitope. Immunogenic peptides whose wild-type counterparts do not elicit immune responses will then be selected for inclusion in an oncolytic virus-based vaccine to be analysed in vivo using transgenic HLA-A2/HLA-DP4 mice [17].

ELIGIBILITY:
Inclusion Criteria:

* fit and healthy;
* weigh over 7 stone 12 lbs or 50kg;
* are aged between 17 and 66 (or 70 if you have given blood before);
* are over 70 and have given blood in the last two years.

Exclusion Criteria:

* receiving treatment;
* taking medication;
* travelling outside of the UK;
* tattoos;
* pregnancy;
* illness;
* cancer;
* received blood, blood products or organs.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy blood donors, who donate their blood at the Blood Donation Centres in London.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2016-09; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Develop Vaccinia virus and Adenovirus vaccine libraries expressing the identified immunogenic neo-epitopes. | 1 month
  To perform in vitro validation of neo-epitope candidates selected from available mutanome data to determine their immunogenicity using peripheral blood mononuclear cells (PBMCs) from healthy individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Cancer Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The research data will be made public on ClinicalTrials.gov.